CLINICAL TRIAL: NCT06851312
Title: Prospective Observational Study to Assess the Implementation of Minimally Invasive Surgery in the Treatment of Grade III Hemorrhoids: Phase 1 of the IDEAL Framework
Brief Title: Implementation of Minimally Invasive Surgery for Grade III Hemorrhoids
Status: Completed | Type: Observational
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Ignacio Fernandez Hurtado, Principal Investigator, Hospital Son Llatzer
Other Study IDs: HEM IDEAL1
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhoidectomy; Minimal Invasive Surgery
Keywords: hemorrhoids grade III-IV; Hemorrhoidectomy; Minimal Invasive Surgery; IDEAl Stage 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Grade III Hemorrhoids: Patients with symptomatic grade III hemorrhoids who consent to surgical intervention
  Interventions: Procedure: Minimal invasive hemorrhoidectomy

INTERVENTIONS:
Procedure: Minimal invasive hemorrhoidectomy — We propose applying minimally invasive surgery in open excisional hemorrhoidectomy, the most effective technique for treating advanced hemorrhoidal disease. We believe this approach will reduce postoperative pain and improve recovery while maintaining the excellent outcomes of OEH. Our hypothesis is based on the reduced tissue trauma and increased precision provided by minimally invasive surgery.

SUMMARY:
Hemorrhoids are vascular-elastic structures of the anal canal that contribute to continence. Their enlargement and descent lead to symptoms such as rectal bleeding and the sensation of anal swelling, known as hemorrhoidal syndrome. In advanced cases (Goligher Grade III-IV), surgery is the only effective treatment. Open excisional hemorrhoidectomy (OEH), based on the Milligan-Morgan technique, is the standard procedure. Although effective in the long term, it causes severe postoperative pain.

Minimally invasive surgery (MIS) employs enhanced visualization devices to improve surgical precision and reduce tissue damage. While widely used in specialties with small surgical fields, it has not yet been explored in anal surgery. Its advantages include reduced tissue injury and improved healing, although it presents a learning curve and an initially longer surgical time.

The IDEAL framework evaluates surgical innovations in five stages: Idea, Development, Exploration, Evaluation, and Long-Term Study. In Stage 1, the first application in humans is documented, analyzing outcomes and feasibility.

Since no previous studies on the application of MIS in OEH have been found, the investigators propose a study within Stage 1 of the IDEAL model to assess the feasibility of this technique. The investigators believe its incorporation into open excisional hemorrhoidectomy could result in less postoperative pain and faster patient recovery.

ELIGIBILITY:
INCLUSION CRITERIA

* Age over 18 years
* Grade III hemorrhoids
* BMI below 30
* Indication for OEH surgery
* Signed written informed consent

EXCLUSION CRITERIA

* Acute hemorrhoidal disease (thrombosis)
* Previous hemorrhoid surgery
* Coexistence of anal fissure
* Coexistence of perianal fistula
* Coexistence of rectal or anal prolapse
* Active inflammatory bowel disease
* Active anal or colorectal cancer
* Language barrier or difficulty in oral and/or written comprehension

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending the Surgery Department of our Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Technical Feasibility of Surgery | From enrollment to the surgical procedure
  Since no studies using this approach were found in the literature, the investigators propose a study to assess the feasibility of implementing this technique following the guidelines of the IDEAL framework. In this study, the investigators propose Stage 1. The measurement tool will be the number of patients in whom the technique could be performed

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Fernandez Hurtado, Colorectal Surgeon, Principal Investigator — Hospital Son Llatzer
Locations (1):
- Hospital Son Llatzer, Palma, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hirst A, Philippou Y, Blazeby J, Campbell B, Campbell M, Feinberg J, Rovers M, Blencowe N, Pennell C, Quinn T, Rogers W, Cook J, Kolias AG, Agha R, Dahm P, Sedrakyan A, McCulloch P. No Surgical Innovation Without Evaluation: Evolution and Further Development of the IDEAL Framework and Recommendations. Ann Surg. 2019 Feb;269(2):211-220. doi: 10.1097/SLA.0000000000002794. PMID 29697448
- [Background] McCulloch P, Altman DG, Campbell WB, Flum DR, Glasziou P, Marshall JC, Nicholl J; Balliol Collaboration; Aronson JK, Barkun JS, Blazeby JM, Boutron IC, Campbell WB, Clavien PA, Cook JA, Ergina PL, Feldman LS, Flum DR, Maddern GJ, Nicholl J, Reeves BC, Seiler CM, Strasberg SM, Meakins JL, Ashby D, Black N, Bunker J, Burton M, Campbell M, Chalkidou K, Chalmers I, de Leval M, Deeks J, Ergina PL, Grant A, Gray M, Greenhalgh R, Jenicek M, Kehoe S, Lilford R, Littlejohns P, Loke Y, Madhock R, McPherson K, Meakins J, Rothwell P, Summerskill B, Taggart D, Tekkis P, Thompson M, Treasure T, Trohler U, Vandenbroucke J. No surgical innovation without evaluation: the IDEAL recommendations. Lancet. 2009 Sep 26;374(9695):1105-12. doi: 10.1016/S0140-6736(09)61116-8. PMID 19782876